CLINICAL TRIAL: NCT06903013
Title: Post Operative Pain Following Pulpectomy Versus Pulpotomy in Primary Molars Wit Irreversible Pulpitis a Parallel Randomized Clinical Trial
Brief Title: Post Operative Pain Following Pulpectomy Versus Pulpotomy in Primary Molars Wit Irreversible Pulpitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mahmoud, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1029
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulpotomy (Experimental): Vital pulpotomy using regenerative materials
  Interventions: Other: Vital pulp therapy
- Pulpectomy (Active Comparator)
  Interventions: Other: Non vitalPulp therapy

INTERVENTIONS:
Other: Non vitalPulp therapy — Pulp therapy deals about management of inflamed vital dental pulp With complete pulp removal and obturation with resorbable materi
  Arms: Pulpectomy
Other: Vital pulp therapy — Pulp therapy through partial root removal and using of regenerative capping material
  Arms: Pulpotomy

SUMMARY:
Study will evaluate and compare post operative pain for primary molars with irreversible pulpitis after pulpotomy and pulpuectomy

ELIGIBILITY:
Inclusion Criteria:

* Healthy individual
* Has primary tooth with irreversible pulpitis
* Cooperative child

Exclusion Criteria:

* Mentally, physically or medically compromised children
* Uncooperative children

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 6 months
  Post operative pain using pain scale after 1,2,7 days